CLINICAL TRIAL: NCT00083551
Title: UARK 98-026, Total Therapy II - A Phase III Study for Newly Diagnosed Multiple Myeloma Evaluating Anti-Angiogenesis With Thalidomide and Post-Transplant Consolidation Chemotherapy
Brief Title: UARK 98-026 TT II: Multiple Myeloma Evaluating Anti-Angiogenesis With Thalidomide and Post-Transplant Consolidation Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5226
Record Dates: First submitted 2004-05-25; First posted 2004-05-27 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; Therapy; Thalidomide; DTPACE; Transplant; VAD; DCEP; CAD; Consolidation; Melphalan
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Thalidomide; Cytarabine; Carmustine; Cisplatin; Cyclophosphamide; Dexamethasone; Tobramycin, Dexamethasone Drug Combination; Doxorubicin; Etoposide; etoposide phosphate; Filgrastim; Introns; Melphalan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide (Active Comparator): Thalidomide 400 qod during induction.100 mg qd between transplants, post transplant pat. 200 mg qd. During year one of maintenance therapy pt will take 100mg of Thal qod and 50 mg of thal qod during second year of maintenance
  Interventions: Drug: Thalidomide; Drug: Ara-C; Drug: BCNU; Drug: Cisplatin; Drug: Cytoxan; Drug: Dexamethasone; Drug: Etoposide; Drug: Filgrastim; Drug: Recombinant GM-CSF; Drug: Interferon-alpha-2b; Drug: Melphalan
- No Thalidomide (Active Comparator): During induction, consolidation, and maintenance steps patient receives no thalidamide
  Interventions: Drug: Ara-C; Drug: BCNU; Drug: Cisplatin; Drug: Cytoxan; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Etoposide; Drug: Filgrastim; Drug: Recombinant GM-CSF; Drug: Interferon-alpha-2b; Drug: Melphalan; Drug: Vincristine

INTERVENTIONS:
Drug: Thalidomide — All patients will be randomly assigned to receive thalidomide 400 mg as an oral, once daily dose throughout induction and 100mg between transplants after platelets are greater than 50,000μl and 200 mg post transplant consolidation, and a reduced dose of 100 mg on alternating days during the first year of maintenance and 50 mg qod thereafter versus no thalidomide. Thalidomide will be held during conditioning, transplant procedure, and recovery following transplant. It may be resumed once plateletrecovery is complete after each transplant
  Other Names: Thalomid
  Arms: Thalidomide
Drug: Ara-C — Cytarabine (Ara-C) 400 mg/m2 in 250 ml D5W over one hour daily for four days (on days -5, -4, -3, -2).
  Start infusion 30 minutes after completion of BCNU on day -5.
  Other Names: Cytarabine
Drug: BCNU — Carmustine (BCNU) 300 mg/m2 in 1 liter of D5W in glass bottle (protect from light) to infuse over 2 hours on day -5. Check blood pressure every 15 minutes during infusion and 30 minutes after completion
  Other Names: Carmustine
Drug: Cisplatin — Cisplatin* 15 mg/m2/day Continuous infusion 1-4 (DCEP CYCLE 2) Cisplatin* 7.5 mg/m2 Continuous infusion 1-4 (DPACE cycle)
  *Cisplatin doses will be modified for renal insufficiency as follows: Cisplatin dose Creatinine 15 mg/m2 (full dose) < 1.5 mg/dl 10 mg/m2 1.6 - 2.0 mg/dl 7.5 mg/m2 2.1 - 3.0 mg/dl 0 mg (hold Cisplatin) > 3.0 mg/dl
  Other Names: cisplatinum; cis-diamminedichloroplatinum; Platinol; Platinol-AQ
Drug: Cytoxan — Cycle 2 - DCEP Cyclophosphamide 400 mg/m2/day Continuous infusion 1-4 Cycle 3 - CAD and PBSC Collection #1 Cyclophosphamide 750 mg/m2/day Continuous infusion 1-4 Cycle 4 - DCEP Cyclophosphamide 400 mg/m2/day Continuous infusion 1-4 Cytoxan/VP-16 and PBSC Collection-Cyclophosphamide 2 grams/m2 (Total dose 4 gm/m2) IV by CI 1 and 2 Post-Transplant Consolidation-Cyclophosphamide 300 mg/m2 Continuous infusion 1-4
  Other Names: Cyclophosphamide; Endoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Dexamethasone — Induction cycle 1 VAD Dexamethasone 40 mg/day PO 1-4, 9-12, 17-20 Cycle 2 - DCEP Dexamethasone 40 mg/day PO 1-4 Cycle 3 - CAD and PBSC Collection #1 Dexamethasone 40 mg/day PO 1-4 Cycle 4 - DCEP and PBSC Collection #2 Dexamethasone 40 mg/day PO 1-4 Post-Transplant Consolidation Dexamethasone 40 mg PO 1-4 Dexamethasone Consolidation Patients that do not achieve adequate platelet recovery (defined as < 80,000/μl) will receive consolidation with Dexamethasone 40 mg x 4 days every 28 days for 1 year Maintenance year one Dexamethasone 40 mg PO q 3 months, day 1-4, 9-12, 17-20
  Other Names: Tobradex
Drug: Doxorubicin — Doxorubicin may be further diluted in 5% dextrose or sodium chloride injection and should be administered slowly into tubing of a freely flowing intravenous infusion with great care taken to avoid extravasation.
  Other Names: Adriamycin; hydroxydaunorubicin
  Arms: No Thalidomide
Drug: Etoposide — Etoposide (VP16) 200 mg/m2 in 500 ml D5W over one hour daily for four days (on days -5, -4, -3, -2). Start infusion 30 minutes after completion of BCNU on day -5. Start infusion at completion of cytarabine on following three days
  Other Names: Eposin; Etopophos; Vepesid; VP-16
Drug: Filgrastim — G-CSF will be administered at a dose of 10mcg/kg or GM-CSF at a dose of 10 mcg/kg. G-CSF or GM-CSF will begin one day after completion of chemotherapy and continued during repeated apheresis and discontinued upon completion of apheresis.
  Other Names: Neupogen; Grafeel; Religrast; Nugraf; Shilgrast; Neukine; Emgrast
Drug: Recombinant GM-CSF — GM-CSF at a dose of 10 μg/kg SC, divided in 2 doses each day, will begin one day after completion of chemotherapy and continued during repeated apheresis and discontinued upon completion of apheresis.
Drug: Interferon-alpha-2b — AGENT DOSE ROUTE DAYS Intron-A 3 million units/m2 SQ TIW Thalidomide (for those randomized at initial registration) 50 mg QOD PO Every other day (qod
Drug: Melphalan — Etoposide (VP16) 200 mg/m2 in 500 ml D5W over one hour daily for four days (on days -5, -4, -3, -2). Start infusion 30 minutes after completion of BCNU on day -5. Start infusion at completion of cytarabine on following three days
  Other Names: Alkeran
Drug: Vincristine — Formulation: 1 mg/1 ml, 2 mg/2 ml, and 5 mg/ 5 ml vials. Vincristine should be administered intravenously through a freely-running IV. If it extravasates, it produces a severe local reaction with skin slough. FATAL IF GIVEN INTRATHECALLY, FOR INTRAVENOUS USE ONLY.
  Other Names: Oncovin; leurocristine
  Arms: No Thalidomide

SUMMARY:
This study has been designed to evaluate whether "anti-angiogenesis" therapy with thalidomide and whether additional chemotherapy after transplant will be beneficial. Another objective is to find out what kinds of side effects occur with this combination of treatment and how often they occur.

DETAILED DESCRIPTION:
Treatment will be given in 4 phases or steps: Induction, Transplant 1 and 2, Consolidation, and maintenance. Induction is designed to induce (or bring about) myeloma into remission. Each patient enrolled on this study will be randomly assigned to receive the above treatment alone or in combination with a drug called thalidomide. Some patients may be eligible to receive the transplant as an outpatient, based on general health and other factors.After recovery from the transplant phase of the study (approximately 6 weeks), patients originally assigned to thalidomide will resume taking it and will continue taking it throughout the rest of the study treatment. All patients will receive post-transplant consolidation treatment, which in earlier studies has been found to be helpful in maintaining patients response after transplant. Therefore, all patients will receive a combination of drugs called "D PACE" which consists of Dexamethasone, Cis-Platinum, Adriamycin, Cyclophosphamide, and Etoposide. If you are also taking thalidomide, you will continue taking it throughout, and the treatment is called "DT PACE" to include the thalidomide. No sooner than 4 weeks, and no later than 12 weeks after consolidation and if your myeloma remains in remission after consolidation therapy is complete, you will begin the last phase of the study, which is maintenance. Maintenance is designed to keep your myeloma in remission long-term.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active multiple myeloma requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Protein criteria must be present in order to evaluate response.Non-secretory patients are eligible provided the patient has > or = 20% plasmacytosis or multiple (>3) focal plasmacytomas on MRI or diffuse hyperintense signal on STIR images in the absence of hematopoietic growth factors is seen.
* All necessary baseline studies for determining stage, bloodwork, and bone marrow must be obtained within 35 days prior to registration.
* Patients must have received no more than one cycle of prior chemotherapy including one month of Dexamethasone and Thalidomide for this disease. Patients may have received prior radiotherapy provided approval has been obtained by one of the study coordinators.
* Patients must have a performance status of 0-2 based on SWOG criteria. Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* Patients with renal failure, even if on dialysis, are eligible if it is felt to be due to myeloma and if the duration of renal failure does not exceed two months
* Patients must be 75 years of age or less at the time of registration
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* If medically appropriate, patients with pathologic fractures, pneumonia at diagnosis or hyperviscosity with shortness of breath should have these conditions attended to prior to registration.

Exclusion Criteria:

* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection
* Patients must not have uncontrolled diabetes
* Patients with recent (< or =6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrythmias are ineligible. Ejection fraction by ECHO or MUGA should be within the institutional normal range and must be performed within 42 days prior to registration.
* Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years.Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval and there must be no prior treatment with cytotoxic drugs that could potentially be assigned on this treatment protocol.
* Pregnant or nursing women may not participate. Women of child-bearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use two forms of effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 1998-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, M.D., Ph.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Barlogie B, Tricot G, Anaissie E, Shaughnessy J, Rasmussen E, van Rhee F, Fassas A, Zangari M, Hollmig K, Pineda-Roman M, Lee C, Talamo G, Thertulien R, Kiwan E, Krishna S, Fox M, Crowley J. Thalidomide and hematopoietic-cell transplantation for multiple myeloma. N Engl J Med. 2006 Mar 9;354(10):1021-30. doi: 10.1056/NEJMoa053583. PMID 16525139
- [Derived] Al Hadidi S, Ababneh OE, Schinke CD, Thanendrarajan S, Siegel ER, Bailey C, Smith R, Panozzo SB, Zangari M, Tricot G, Shaughnessy JD Jr, Zhan F, Sawyer J, Barlogie B, van Rhee F. Long-Term Follow-Up of Patients With Multiple Myeloma Treated on Earlier Total Therapy Protocols: A Secondary Analysis of 3 Clinical Trials. JAMA Oncol. 2025 Aug 1;11(8):910-915. doi: 10.1001/jamaoncol.2025.1394. PMID 40471585
- [Derived] Vatsveen TK, Sponaas AM, Tian E, Zhang Q, Misund K, Sundan A, Borset M, Waage A, Brede G. Erythropoietin (EPO)-receptor signaling induces cell death of primary myeloma cells in vitro. J Hematol Oncol. 2016 Aug 31;9(1):75. doi: 10.1186/s13045-016-0306-x. PMID 27581518
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Thalidomide: Thalidomide 400 QD during induction, 100 mg QD between transplants, 200 mg QD post transplant, 100 mg QD during year one of maintenance, and 50 mg QD during second year of maintenance.
- No Thalidomide: Patient received no thalidomide during induction, consolidation, and maintenance therapy.
Period: Overall Study
Arm/Group | Thalidomide | No Thalidomide
Started | 323 | 345
Completed | 323 | 345
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thalidomide | No Thalidomide | Total
Number analyzed (Participants) | 323 | 345 | 668
Age, Customized [Number; unit: participants]
  >/= 60 to < 65 years | 130 | 129 | 259
  >/= 65 years | 64 | 72 | 136
  < 60 years | 129 | 144 | 273
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 135 | 272
  Male | 186 | 210 | 396

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival at six years after initiating protocol therapy
Time Frame: 6 Years
Measure: Number; unit: percentage of participants
Arm/Group | Thalidomide | No Thalidomide
Number analyzed (Participants) | 323 | 345
percentage of participants | 65 | 58

ADVERSE EVENTS:
Arm/Group | Thalidomide | No Thalidomide
Serious Adverse Events (participants affected / at risk) | 323/323 | 345/345
Other Adverse Events (participants affected / at risk) | 323/323 | 345/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide (N=323) | No Thalidomide (N=345)
Grade 3 Arrhythmia, NOS (Cardiac disorders) | 12 | 21
Grade 4 Arrhythmia, NOS (Cardiac disorders) | 2 | 2
Grade 3 Cardiac ischemia/infarction (Cardiac disorders) | 3 | 2
Grade 4 Cardiac ischemia/infarction (Cardiac disorders) | 2 | 1
Grade 3 Cardiovascular-other (Cardiac disorders) | 7 | 1
Grade 4 Cardiovascular-other (Cardiac disorders) | 0 | 1
Grade 3 Cerebrovascular ischemia (Cardiac disorders) | 7 | 2
Grade 4 Cerebrovascular ischemia (Cardiac disorders) | 1 | 0
Grade 3 Conduction abnormality/block (Cardiac disorders) | 0 | 1
Grade 4 Conduction abnormality/block (Cardiac disorders) | 0 | 1
Grade 3 Edema (Cardiac disorders) | 6 | 4
Grade 3 Hypertension (Cardiac disorders) | 7 | 7
Grade 3 Hypotension (Cardiac disorders) | 8 | 8
Grade 4 Hypotension (Cardiac disorders) | 5 | 0
Grade 3 LVEF decrease/CHF (Cardiac disorders) | 0 | 2
Grade 3 Nodal/junctional dysrhythmia (Cardiac disorders) | 1 | 0
Grade 3 Sinus bradycardia (Cardiac disorders) | 6 | 2
Grade 4 Sinus bradycardia (Cardiac disorders) | 1 | 0
Grade 3 Sinus tachycardia (Cardiac disorders) | 3 | 2
Grade 3 Supraventricular arrhythmia (Cardiac disorders) | 7 | 7
Grade 4 Supraventricular arrhythmia (Cardiac disorders) | 0 | 1
Grade 3 Surgery-injury of vein/artery (Cardiac disorders) | 0 | 1
Grade 3 Syncope (Cardiac disorders) | 31 | 12
Grade 3 Thrombosis/embolism (Cardiac disorders) | 69 | 47
Grade 4 Thrombosis/embolism (Cardiac disorders) | 11 | 3
Grade 3 Valvular heart disease (Cardiac disorders) | 1 | 0
Grade 3 Vasovagal episode (Cardiac disorders) | 1 | 0
Grade 3 Ventricular arrhythmia (Cardiac disorders) | 2 | 3
Grade 4 Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Grade 3 Supra Arrhyth: Atrial Fib. (Cardiac disorders) | 1 | 0
Grade 3 Clotting-other (Blood and lymphatic system disorders) | 1 | 0
Grade 3 Prothrombin time increase (Blood and lymphatic system disorders) | 1 | 0
Grade 3 Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Grade 3 Hearing (Ear and labyrinth disorders) | 1 | 1
Grade 3 Inner ear - hearing loss (Ear and labyrinth disorders) | 8 | 0
Grade 3 Middle ear - hearing loss/otitis (Ear and labyrinth disorders) | 2 | 1
Grade 3 Diabetes (Endocrine disorders) | 1 | 1
Grade 3 Endocrine - other (Endocrine disorders) | 1 | 0
Grade 3 SIADH (Endocrine disorders) | 0 | 1
Grade 3 Blurred vision (Eye disorders) | 3 | 2
Grade 3 Cataract (Eye disorders) | 10 | 4
Grade 3 Double vision (Eye disorders) | 0 | 1
Grade 3 Eye - other (Eye disorders) | 2 | 1
Grade 3 Keratitis (Eye disorders) | 0 | 1
Grade 3 Photophobia (Eye disorders) | 0 | 1
Grade 4 Retinopathy (Eye disorders) | 1 | 0
Grade 3 Fatigue/malaise/lethargy (General disorders) | 130 | 139
Grade 4 Fatigue/malaise/lethargy (General disorders) | 40 | 52
Grade 3 Fever without neutropenia (General disorders) | 2 | 8
Grade 4 Fever without neutropenia (General disorders) | 0 | 1
Grade 3 Fever, NOS (General disorders) | 29 | 25
Grade 4 Fever, NOS (General disorders) | 2 | 3
Grade 3 Flu-like symptoms-other (General disorders) | 3 | 4
Grade 3 Insomnia (General disorders) | 1 | 0
Grade 3 Obesity (General disorders) | 0 | 1
Grade 3 Rigors/chills (General disorders) | 0 | 1
Grade 4 Sweating (General disorders) | 0 | 1
Grade 3 Weight loss (General disorders) | 1 | 1
Grade 3 Anal incontinence (Gastrointestinal disorders) | 1 | 0
Grade 3 Anorexia (Gastrointestinal disorders) | 94 | 99
Grade 4 Anorexia (Gastrointestinal disorders) | 6 | 6
Grade 3 Colitis (Gastrointestinal disorders) | 8 | 5
Grade 4 Colitis (Gastrointestinal disorders) | 1 | 7
Grade 3 Constipation/bowel obstruction (Gastrointestinal disorders) | 31 | 17
Grade 4 Constipation/bowel obstruction (Gastrointestinal disorders) | 6 | 8
Grade 3 Dehydration (Gastrointestinal disorders) | 4 | 5
Grade 3 Diarrhea with colostomy (Gastrointestinal disorders) | 1 | 4
Grade 3 Diarrhea without colostomy (Gastrointestinal disorders) | 61 | 80
Grade 4 Diarrhea without colostomy (Gastrointestinal disorders) | 8 | 7
Grade 3 Dyspepsia/heartburn (Gastrointestinal disorders) | 3 | 2
Grade 3 Esophagitis/dysphagia (Gastrointestinal disorders) | 26 | 35
Grade 4 Esophagitis/dysphagia (Gastrointestinal disorders) | 10 | 7
Grade 3 Dysphagia (Gastrointestinal disorders) | 1 | 0
Grade 3 GI Mucositis, NOS (Gastrointestinal disorders) | 20 | 10
Grade 4 GI Mucositis, NOS (Gastrointestinal disorders) | 0 | 1
Grade 3 GI-other (Gastrointestinal disorders) | 2 | 6
Grade 4 GI-other (Gastrointestinal disorders) | 2 | 1
Grade 3 Ileus (Gastrointestinal disorders) | 0 | 2
Grade 3 Mouth Dryness (Gastrointestinal disorders) | 7 | 5
Grade 4 Mouth Dryness (Gastrointestinal disorders) | 0 | 1
Grade 3 Nausea (Gastrointestinal disorders) | 117 | 118
Grade 4 Nausea (Gastrointestinal disorders) | 3 | 4
Grade 3 Pancreatitis (Gastrointestinal disorders) | 1 | 0
Grade 3 Periodontal (Gastrointestinal disorders) | 1 | 0
Grade 3 RT-GI mucositis, NOS (Gastrointestinal disorders) | 1 | 0
Grade 3 Stomatitis/pharyngitis (Gastrointestinal disorders) | 60 | 41
Grade 4 Stomatitis/pharyngitis (Gastrointestinal disorders) | 7 | 12
Grade 3 Vomiting (Gastrointestinal disorders) | 37 | 42
Grade 4 Vomiting (Gastrointestinal disorders) | 6 | 8
Grade 3 Bladder Spasms (Renal and urinary disorders) | 4 | 2
Grade 4 Bladder Spasms (Renal and urinary disorders) | 1 | 1
Grade 3 Creatinine increase (Renal and urinary disorders) | 12 | 8
Grade 4 Creatinine increase (Renal and urinary disorders) | 16 | 15
Grade 3 GU-other (Renal and urinary disorders) | 2 | 1
Grade 3 incontinence (Renal and urinary disorders) | 0 | 1
Grade 3 Renal failure (Renal and urinary disorders) | 6 | 6
Grade 4 Renal failure (Renal and urinary disorders) | 8 | 5
Grade 3 Urinary frequency/urgency (Renal and urinary disorders) | 0 | 2
Grade 3 Urinary retention (Renal and urinary disorders) | 1 | 0
Grade 4 Anemia (HGB) (Blood and lymphatic system disorders) | 27 | 34
Grade 4 Neutropenia/granulocytopenia (Blood and lymphatic system disorders) | 242 | 259
Grade 4 Platelet transfusion (Blood and lymphatic system disorders) | 1 | 0
Grade 4 Thrombocytopenia (PLT) (Blood and lymphatic system disorders) | 159 | 168
Grade 4 Leukopenia (WBC) (Blood and lymphatic system disorders) | 257 | 279
Grade 3 Hematuria (Blood and lymphatic system disorders) | 5 | 4
Grade 4 Hematuria (Blood and lymphatic system disorders) | 0 | 1
Grade 3 Hemorrhage w/3-4 thrombocytopenia (Blood and lymphatic system disorders) | 38 | 37
Grade 4 Hemorrhage w/3-4 thrombocytopenia (Blood and lymphatic system disorders) | 6 | 10
Grade 3 Hemorrhage w/o 3-4 thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Grade 3 Hemorrhage-other (Blood and lymphatic system disorders) | 1 | 0
Grade 4 Vaginal bleeding (Blood and lymphatic system disorders) | 1 | 0
Grade 3 Petechiae/purpura (Blood and lymphatic system disorders) | 0 | 1
Grade 3 Melena/GI bleeding (Blood and lymphatic system disorders) | 6 | 9
Grade 4 Melena/GI bleeding (Blood and lymphatic system disorders) | 2 | 2
Grade 3 Allergic/hypersensitivity (Immune system disorders) | 0 | 1
Grade 3 Autoimmune reaction (Immune system disorders) | 4 | 1
Grade 4 Autoimmune reaction (Immune system disorders) | 4 | 0
Grade 3 Catheter related infection (Infections and infestations) | 11 | 18
Grade 3 Ear infection ANC mid ear (Infections and infestations) | 0 | 1
Grade 3 Febrile neutropenia (Infections and infestations) | 62 | 80
Grade 4 Febrile neutropenia (Infections and infestations) | 0 | 2
Grade 3 GI infection 3-4 ANC abdomen (Infections and infestations) | 0 | 1
Grade 3 GI infection 3-4 ANC appendix (Infections and infestations) | 0 | 1
Grade 3 GI Infection 3-4 ANC tooth (Infections and infestations) | 0 | 1
Grade 3 GI infection ANC abdomen (Infections and infestations) | 0 | 1
Grade 3 GU infection ABC UTI (Infections and infestations) | 1 | 0
Grade 3 Infection w/grade 3 or 4 Neutrophils (Infections and infestations) | 3 | 1
Grade 3 Infection w/o 3-4 Neutropenia (Infections and infestations) | 29 | 38
Grade 4 Infection w/o 3-4 Neutropenia (Infections and infestations) | 1 | 1
Grade 3 Infection w/3-4 Neutropenia (Infections and infestations) | 28 | 27
Grade 4 Infection w/3-4 Neutropenia (Infections and infestations) | 0 | 1
Grade 3 Infection ANC (Infections and infestations) | 27 | 25
Grade 4 Infection ANC (Infections and infestations) | 1 | 0
Grade 3 Lung infection 3-4 ANC (Infections and infestations) | 1 | 0
Grade 3 Lung Infection ANC Bronchus (Infections and infestations) | 1 | 0
Grade 3 Lung Infection ANC Lung (Infections and infestations) | 1 | 0
Grade 3 Lung Infection ANC Pharynx (Infections and infestations) | 1 | 0
Grade 3 Moderate (Infections and infestations) | 1 | 2
Grade 3 Respiratory infect w/neutrop (Infections and infestations) | 4 | 2
Grade 3 Muscle infection ANC Bone (Infections and infestations) | 1 | 0
Grade 3 Respiratory infection w/o neutrop (Infections and infestations) | 17 | 10
Grade 4 Respiratory infection w/o neutrop (Infections and infestations) | 1 | 1
Grade 3 Respiratory infection ANC (Infections and infestations) | 18 | 11
Grade 3 Skin infection 3-4 ANC lip/perior (Infections and infestations) | 1 | 0
Grade 3 Surgery-wound infection (Infections and infestations) | 2 | 0
Grade 4 Surgery -wound infection (Infections and infestations) | 1 | 0
Grade 3 Urinary tract infectiob w/neutrop (Infections and infestations) | 0 | 1
Grade 3 Uninary tract infection w/o neutrop (Infections and infestations) | 1 | 2
Grade 4 Urinary tract infection w/o neutrop (Infections and infestations) | 0 | 1
Grade 3 Urinary tract infection ANC (Infections and infestations) | 2 | 3
Grade 3 Alkaline phosphatase increase (Hepatobiliary disorders) | 3 | 4
Grade 3 Bilirubin increase (Hepatobiliary disorders) | 8 | 9
Grade 4 Bilirnbin increase (Hepatobiliary disorders) | 4 | 2
Grade 3 Hypoalbuminemia (Hepatobiliary disorders) | 16 | 18
Grade 3 Liver enlargement (Hepatobiliary disorders) | 0 | 1
Grade 3 SGOT (AST) increase (Hepatobiliary disorders) | 9 | 7
Grade 4 SGOT (AST) increase (Hepatobiliary disorders) | 0 | 3
Grade 3 SGPT (ALT) increase (Hepatobiliary disorders) | 18 | 19
Grade 4 SGPT (ALT) increase (Hepatobiliary disorders) | 1 | 1
Grade 4 Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Grade 3 Apnea (Nervous system disorders) | 2 | 0
Grade 4 Apnea (Nervous system disorders) | 1 | 0
Grade 3 Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 12
Grade 4 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Grade 3 Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Grade 3 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 33 | 37
Grade 4 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Grade 3 Lung Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Grade 3 Lung-other (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Grade 4 Lung-other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Grade 3 Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Grade 3 Pneumonitis/infilitrates (Respiratory, thoracic and mediastinal disorders) | 35 | 30
Grade 4 Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Grade 3 Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Grade 3 Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Grade 3 Voice charge /stridor/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Grade 3 Bicarbonate decrease (Metabolism and nutrition disorders) | 8 | 5
Grade 4 Bicarbonate decrease (Metabolism and nutrition disorders) | 1 | 1
Grade 3 Hypercalcemia (Metabolism and nutrition disorders) | 2 | 4
Grade 4 Hypercalcemia (Metabolism and nutrition disorders) | 6 | 2
Grade 3 Hyperglycemia (Metabolism and nutrition disorders) | 57 | 84
Grade 4 Hyperglycemia (Metabolism and nutrition disorders) | 10 | 10
Grade 3 Hyperkalemia (Metabolism and nutrition disorders) | 11 | 18
Grade 4 Hyperkalemia (Metabolism and nutrition disorders) | 5 | 3
Grade 3 Hypermagnesemia (Metabolism and nutrition disorders) | 14 | 21
Grade 4 Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Grade 3 Hypermatremia (Metabolism and nutrition disorders) | 0 | 2
Grade 4 Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Grade 3 Hypocalcemia (Metabolism and nutrition disorders) | 61 | 75
Grade 4 Hypocalcemia (Metabolism and nutrition disorders) | 20 | 17
Grade 3 Hypokalemia (Metabolism and nutrition disorders) | 72 | 89
Grade 4 Hypokalemia (Metabolism and nutrition disorders) | 6 | 3
Grade 3 Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 10
Grade 4 Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 101 | 95
Grade 4 Hyponatremia (Metabolism and nutrition disorders) | 14 | 8
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 183 | 214
Grade 4 Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Grade 3 Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Grade 2 Gait/Walking (Musculoskeletal and connective tissue disorders) | 3 | 0
Grade 4 Gait/Walking (Musculoskeletal and connective tissue disorders) | 1 | 0
Grade 3 Joint, muscle, bone (Musculoskeletal and connective tissue disorders) | 19 | 6
Grade 3 Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 5
Grade 3 Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Grade 3 Anxiety/agitation (Nervous system disorders) | 8 | 16
Grade 4 Anxiety/agitation (Nervous system disorders) | 3 | 5
Grade 3 Ataxia (Nervous system disorders) | 10 | 6
Grade 4 CNS ischemia (Nervous system disorders) | 1 | 0
Grade 3 Confusion (Nervous system disorders) | 25 | 23
Grade 4 Confusion (Nervous system disorders) | 5 | 8
Grade 3 Depression (Nervous system disorders) | 32 | 28
Grade 4 Depression (Nervous system disorders) | 6 | 6
Grade 3 Dizziness/light headedness (Nervous system disorders) | 35 | 15
Grade 4 Dizziness/light headedness (Nervous system disorders) | 4 | 3
Grade 3 Dizziness/vertigo (Nervous system disorders) | 1 | 0
Grade 3 Hallucinations (Nervous system disorders) | 4 | 2
Grade 3 Headache (Nervous system disorders) | 11 | 19
Grade 3 Insomnia (Nervous system disorders) | 4 | 4
Grade 3 Involuntary movement/restlessnes (Nervous system disorders) | 1 | 0
Grade 3 Mood/consciousness change (Nervous system disorders) | 23 | 17
Grade 4 Mood/consciousness change (Nervous system disorders) | 2 | 3
Grade 3 Neuro-other (Nervous system disorders) | 3 | 3
Grade 4 Neuro-other (Nervous system disorders) | 0 | 1
Grade 3 Seizures (Nervous system disorders) | 2 | 1
Grade 4 Seizures (Nervous system disorders) | 0 | 3
Grade 3 Sensory/neuropathy (Nervous system disorders) | 46 | 13
Grade 4 Sensory/neuropathy (Nervous system disorders) | 1 | 0
Grade 3 Somnolence/consciousness loss (Nervous system disorders) | 40 | 32
Grade 4 Somnolence/consciousness loss (Nervous system disorders) | 4 | 4
Grade 3 Speech impairment (Nervous system disorders) | 0 | 1
Grade 3 Tremor (Nervous system disorders) | 32 | 15
Grade4 Tremor (Nervous system disorders) | 2 | 1
Grade 3 Weakness (motor neuropathy) (Nervous system disorders) | 55 | 36
Grade 4 Weakness (motor neuropathy) (Nervous system disorders) | 3 | 5
Grade 3 Abdominal pain/cramping (General disorders) | 10 | 8
Grade 4 Abdominal pain/cramping (General disorders) | 0 | 1
Grade 3 Arthralgia (General disorders) | 6 | 8
Grade 4 Arthralgia (General disorders) | 0 | 1
Grade 3 Bone pain (General disorders) | 24 | 18
Grade 4 Bone pain (General disorders) | 4 | 4
Grade 3 Cardiac/heart (Cardiac disorders) | 1 | 0
Grade 3 Chest/thorax (Cardiac disorders) | 0 | 1
Grade 3 Chest pain/not cardio or pleural (General disorders) | 2 | 4
Grade 3 Earache (Ear and labyrinth disorders) | 2 | 0
Grade 3 Extremity/limb (General disorders) | 1 | 2
Grade 3 Eye (Eye disorders) | 0 | 1
Grade 3 Hepatic pain (General disorders) | 0 | 1
Grade 3 Hip-left (General disorders) | 1 | 0
Grade 3 Lower back (General disorders) | 1 | 3
Grade 3 Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Grade 3 Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Grade 3 Myalgia/arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Grade 3 Neuropathic pain (General disorders) | 0 | 3
Grade 3 Pain NOS (General disorders) | 0 | 1
Grade 3 Pain/other (General disorders) | 53 | 47
Grade 4 Pain/other (General disorders) | 4 | 0
Grade 3 Pelvic (General disorders) | 0 | 1
Grade 3 Pleuritic pain (General disorders) | 2 | 0
Grade 3 Rectal/perirectal pain (General disorders) | 1 | 1
Grade 3 Rib (General disorders) | 0 | 1
Grade 3 Tumor pain (General disorders) | 0 | 1
Grade 3 Upper Back (General disorders) | 6 | 4
Grade 4 Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Grade 3 Erectile impotence (Reproductive system and breast disorders) | 1 | 0
Grade 3 Female sterility (Reproductive system and breast disorders) | 1 | 0
Grade 3 Menses changes (Reproductive system and breast disorders) | 1 | 0
Grade 3 Decubitus (Skin and subcutaneous tissue disorders) | 1 | 0
Grade 3 Erythema multifrme/blistering (Skin and subcutaneous tissue disorders) | 1 | 0
Grade 3 Erythema/rash/eruption/desquamation (Skin and subcutaneous tissue disorders) | 6 | 6
Grade 3 Pruritis (Skin and subcutaneous tissue disorders) | 1 | 2
Grade 3 Rash/desquamation (Skin and subcutaneous tissue disorders) | 34 | 36
Grade 4 Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 | 5
Grade 3 Skin/other (Skin and subcutaneous tissue disorders) | 4 | 4
Grade 3 Failure to engraft (General disorders) | 1 | 2
Grade 3 Stem cell infusion complication (General disorders) | 0 | 2
Grade 4 Stem cell infusion complication (General disorders) | 1 | 2
Grade 3 Syndrome/other (General disorders) | 1 | 0
Grade 3 Thrombosis/embolism (General disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide (N=323) | No Thalidomide (N=345)
Grade 1 Arrythmia, NOS (Cardiac disorders) | 70 | 88
Grade 2 Arrythmia, NOS (Cardiac disorders) | 21 | 29
Grade 1 Edema (Cardiac disorders) | 101 | 83
Grade 2 Edema (Cardiac disorders) | 33 | 28
Grade 1 Sinus tachycardia (Cardiac disorders) | 0 | 16
Grade 2 Thrombosis/embolism (Cardiac disorders) | 17 | 21
Grade 1 Hypothyroidism (Endocrine disorders) | 22 | 21
Grade 2 Hypothyroidism (Endocrine disorders) | 30 | 0
Grade 2 Blurred vision (Eye disorders) | 53 | 47
Grade 1 Eye - other (Eye disorders) | 24 | 0
Grade 1 Vision, NOS (Eye disorders) | 16 | 0
Grade 2 Fatigue/malaise/lethargy (General disorders) | 79 | 76
Grade 1 Fever without neutropenia (General disorders) | 48 | 45
Grade 2 Fever without neutropenia (General disorders) | 32 | 21
Grade 1 Fever, NOS (General disorders) | 94 | 112
Grade 2 Fever, NOS (General disorders) | 72 | 59
Grade 1 Flu-like symptoms-other (General disorders) | 35 | 27
Grade 1 Insomnia (General disorders) | 21 | 0
Grade 1 Rigors/chills (General disorders) | 29 | 14
Grade 1 sweating (General disorders) | 37 | 31
Grade 2 sweating (General disorders) | 34 | 36
Grade 1 Weight gain (General disorders) | 36 | 31
Grade 1 Weight loss (General disorders) | 35 | 37
Grade 1 Anorexia (Gastrointestinal disorders) | 50 | 62
Grade 2 Anorexia (Gastrointestinal disorders) | 42 | 44
Grade 2 Colitis (Gastrointestinal disorders) | 0 | 24
Grade 1 Constipation/bowel obstruction (Gastrointestinal disorders) | 55 | 69
Grade 2 Constipation/bowel obstruction (Gastrointestinal disorders) | 143 | 112
Grade 1 Diarrhea without colostomy (Gastrointestinal disorders) | 50 | 51
Grade 2 Diarrhea without colostomy (Gastrointestinal disorders) | 119 | 127
Grade 1 Dyspepsia/heartburn (Gastrointestinal disorders) | 27 | 19
Grade 1 Esophagitis/dysphagia (Gastrointestinal disorders) | 70 | 56
Grade 2 Esophagitis/dysphagia (Gastrointestinal disorders) | 54 | 81
Grade 1 Mouth Dryness (Gastrointestinal disorders) | 52 | 46
Grade 2 Mouth Dryness (Gastrointestinal disorders) | 73 | 48
Grade 1 Nausea (Gastrointestinal disorders) | 46 | 37
Grade 2 Nausea (Gastrointestinal disorders) | 83 | 118
Grade 1 Stomatitis/pharyngitis (Gastrointestinal disorders) | 63 | 66
Grade 2 Stomatitis/pharyngitis (Gastrointestinal disorders) | 73 | 90
Grade 1 Taste Disturbance (Gastrointestinal disorders) | 0 | 17
Grade 1 Vomiting (Gastrointestinal disorders) | 58 | 65
Grade 2 Vomiting (Gastrointestinal disorders) | 105 | 122
Grade 1 Bladder Spasms (Renal and urinary disorders) | 0 | 21
Grade 1 Creatinine increase (Renal and urinary disorders) | 77 | 91
Grade 2 Creatinine increase (Renal and urinary disorders) | 53 | 62
Grade 1 Urinary frequency/urgency (Renal and urinary disorders) | 32 | 22
Grade 2 Anemia (HGB) (Blood and lymphatic system disorders) | 70 | 76
Grade 3 Anemia (HGB) (Blood and lymphatic system disorders) | 161 | 174
Grade 3 Neutropenia/ granulocytopenia (Blood and lymphatic system disorders) | 16 | 20
Grade 3 PRBC transfusion (Blood and lymphatic system disorders) | 25 | 0
Grade 3 Platelet Transfusion (Blood and lymphatic system disorders) | 16 | 0
Grade 3 Thrombocytopenia (PLT) (Blood and lymphatic system disorders) | 99 | 112
Grade 2 Hematuria (Blood and lymphatic system disorders) | 0 | 16
Grade 1 Hemorrhage w/3-4 thrombocytopenia (Blood and lymphatic system disorders) | 40 | 63
Grade 1 Allergic rhinitis (Immune system disorders) | 54 | 42
Grade 1 Autoimmune reaction (Immune system disorders) | 25 | 28
Grade 2 Infection w/Grade 3 or 4 Neutrophils (Infections and infestations) | 21 | 0
Grade 2 Infection w/o 3-4 Neutropenia (Infections and infestations) | 34 | 33
Grade 2 Lung Infection ANC Bronchus (Infections and infestations) | 20 | 15
Grade 2 Respiratory infection w/o neutrop (Infections and infestations) | 33 | 46
Grade 1 Respiratory infection w/o neutrop (Infections and infestations) | 17 | 0
Grade 1 Alkaline phosphatase increase (Hepatobiliary disorders) | 139 | 149
Grade 2 Alkaline phosphatase increase (Hepatobiliary disorders) | 17 | 21
Grade 1 Bilirubin increase (Hepatobiliary disorders) | 52 | 62
Grade 2 Bilirubin increase (Hepatobiliary disorders) | 28 | 24
Grade 1 Hypoalbuminemia (Hepatobiliary disorders) | 86 | 93
Grade 2 Hypoalbuminemia (Hepatobiliary disorders) | 155 | 179
Grade 1 SGOT (AST) increase (Hepatobiliary disorders) | 111 | 124
Grade 2 SGOT (AST) increase (Hepatobiliary disorders) | 25 | 30
Grade 1 SGPT (ALT) increase (Hepatobiliary disorders) | 131 | 140
Grade 2 SGPT (ALT) increase (Hepatobiliary disorders) | 39 | 57
Grade 1 Cough (Respiratory, thoracic and mediastinal disorders) | 113 | 103
Grade 2 Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 31
Grade 2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 97 | 92
Grade 2 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 24 | 24
Grade 2 Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 20 | 22
Grade 1 Edema-limb (General disorders) | 22 | 0
Grade 1 Lymphedema (General disorders) | 16 | 0
Grade 1 Bicarbonate decrease (Metabolism and nutrition disorders) | 194 | 217
Grade 2 Bicarbonate decrease (Metabolism and nutrition disorders) | 28 | 41
Grade 1 Hypercalcemia (Metabolism and nutrition disorders) | 34 | 37
Grade 1 Hyperglycemia (Metabolism and nutrition disorders) | 48 | 48
Grade 2 Hyperglycemia (Metabolism and nutrition disorders) | 152 | 151
Grade 1 Hyperkalemia (Metabolism and nutrition disorders) | 78 | 82
Grade 2 Hyperkalemia (Metabolism and nutrition disorders) | 29 | 15
Grade 1 Hypermagnesemia (Metabolism and nutrition disorders) | 60 | 52
Grade 1 Hypematremia (Metabolism and nutrition disorders) | 80 | 74
Grade 1 Hypocalcemia (Metabolism and nutrition disorders) | 35 | 41
Grade 2 Hypocalcemia (Metabolism and nutrition disorders) | 146 | 160
Grade 1 Hypokalemia (Metabolism and nutrition disorders) | 175 | 182
Grade 1 Hypomagnesemia (Metabolism and nutrition disorders) | 142 | 158
Grade 2 Hypomagnesemia (Metabolism and nutrition disorders) | 119 | 116
Grade 1 Hyponatremia (Metabolism and nutrition disorders) | 141 | 179
Grade 2 Hypophosphatemia (Metabolism and nutrition disorders) | 75 | 65
Grade 1 Joint, muscle, bone (Metabolism and nutrition disorders) | 44 | 40
Grade 2 Joint, muscle, bone (Musculoskeletal and connective tissue disorders) | 22 | 0
Grade 1 Muscle weakness (Musculoskeletal and connective tissue disorders) | 34 | 22
Grade 2 Muscle weakness (Musculoskeletal and connective tissue disorders) | 13 | 20
Grade 1 Anxiety/agitation (Nervous system disorders) | 79 | 93
Grade 2 Anxiety/agitation (Nervous system disorders) | 55 | 44
Grade 1 Ataxia (Nervous system disorders) | 45 | 27
Grade 2 Ataxia (Nervous system disorders) | 27 | 0
Grade 1 Confusion (Nervous system disorders) | 84 | 92
Grade 2 Confusion (Nervous system disorders) | 42 | 35
Grade 1 Depression (Nervous system disorders) | 85 | 101
Grade 2 Depression (Nervous system disorders) | 89 | 94
Grade 1 Dizziness/light headedness (Nervous system disorders) | 76 | 76
Grade 2 Dizziness/light headedness (Nervous system disorders) | 53 | 41
Grade 1 Headache (Nervous system disorders) | 48 | 51
Grade 2 Headache (Nervous system disorders) | 37 | 29
Grade 1 Insomnia (Nervous system disorders) | 46 | 42
Grade 2 Insomnia (Nervous system disorders) | 15 | 0
Grade 1 Memory loss (Nervous system disorders) | 20 | 0
Grade 1 Mood/consciousness change (Nervous system disorders) | 51 | 36
Grade 2 Mood/consciousness change (Nervous system disorders) | 35 | 31
Grade 1 Sensory neuropathy (Nervous system disorders) | 72 | 134
Grade 2 Sensory/neuropathy (Nervous system disorders) | 115 | 62
Grade 1 Somnolence/consciousness loss (Nervous system disorders) | 75 | 78
Grade 2 Somnolence/consciousness loss (Nervous system disorders) | 52 | 34
Grade 1 Tremor (Nervous system disorders) | 64 | 51
Grade 2 Tremor (Nervous system disorders) | 45 | 32
Grade 1 Weakness (motor neuropathy) (Nervous system disorders) | 45 | 52
Grade 2 Weakness (motor neuropathy) (Nervous system disorders) | 77 | 54
Grade 1 Abdominal pain/cramping (General disorders) | 20 | 26
Grade 1 Arthralgia (General disorders) | 60 | 59
Grade 2 Arthralgia (General disorders) | 23 | 27
Grade 1 Bone pain (General disorders) | 77 | 70
Grade 2 Bone pain (General disorders) | 55 | 65
Grade 1 Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 53
Grade 2 Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 14
Grade 1 Pain/other (General disorders) | 53 | 77
Grade 2 Pain/other (General disorders) | 74 | 62
Grade 1 Upper back (General disorders) | 40 | 27
Grade 2 Upper back (General disorders) | 35 | 19
Grade 2 Alopecia (Skin and subcutaneous tissue disorders) | 73 | 79
Grade 1 Bruising (Skin and subcutaneous tissue disorders) | 25 | 27
Grade 1 Dry skin (Skin and subcutaneous tissue disorders) | 60 | 43
Grade 2 Dry skin (Skin and subcutaneous tissue disorders) | 19 | 0
Erythema/rash/eruption/desquamation (Skin and subcutaneous tissue disorders) | 37 | 37
Grade 2 Erythema/rash/eruption/desquamation (Skin and subcutaneous tissue disorders) | 18 | 12
Grade 1 Rash/desquamation (Skin and subcutaneous tissue disorders) | 73 | 86
Grade 2 Rash/desquamation (Skin and subcutaneous tissue disorders) | 82 | 93
Grade 4 Skin/other (Skin and subcutaneous tissue disorders) | 21 | 17
Grade 1 Stem cell infusion complication (General disorders) | 0 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes